CLINICAL TRIAL: NCT01155804
Title: Assessment of the Effectiveness of a Program of Preparation to Pregnancy and Delivery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Research on Reproductive Health of Campinas (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Maria Y. Makuch, Ph.D., Cemicamp
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FAPESP2010
Record Dates: First submitted 2010-06-23; First posted 2010-07-02 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2010-04

CONDITIONS: Lumbago; Anxiety
Keywords: preparation of the delivery; lumbago; anxiety; urinary incontinence
MeSH Terms: conditions — Low Back Pain; Anxiety Disorders; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercice (Other)
  Interventions: Behavioral: preparation of the delivery
- non-exercice (Other)
  Interventions: Behavioral: preparation of the delivery

INTERVENTIONS:
Behavioral: preparation of the delivery — Pregnant nulliparous women allocated to the non-interventional group will follow the routine pre-natal care. The participants of the study group will receive routine attention at the pre-natal care service and will also participate in the program of physical and educational after each routine pre-natal consultation. These activities will be organize as follow: 30 minutes of physical exercise for the prevention of pain and discomfort that may occur during pregnancy, preparation of the perineal muscles for delivery and prevention of urinary incontinence, 15 minutes for relaxation and 30 minutes for group discussion to respond to doubts that women may have and issues such as: change in posture during pregnancy and prevention of pain and discomfort; role of the perineal muscles during pregnancy, delivery and puerperium, physiology of delivery, non-pharmacological way for pain relief and breathing control during contractions of labor and delivery.

SUMMARY:
Introduction: randomized studies on programs implemented during pre-natal care that offer information and physical activities preparing pregnant women for delivery are scarce in the scientific literature. Objective: to evaluate the effectively of the Program for Preparation of Pregnant Women for Delivery on the prevention of physical and psychological difficulties and problems during pregnancy and delivery in nulliparous women participating in the program. Subjects and methods: a randomized clinical single blind trial will be conducted with 192 pregnant nulliparous women allocated to participate or not of the program activities. The women allocated to the study group will participate of physical and educational activities at each pre-natal consultation and will receive orientation on the exercises they will perform at their home. Participants of the non-interventional group will follow the habitual routine care at the service. Participants will be selected among nulliparous low risk pregnant women aged between 16 and 40 years old after the 20th week of gestation. Data analysis: will be performing by intention to treat. For the continues variables the t-Student or Wilcoxon test will be performing; for the categorical variables the tests x² or Fisher, and the risk estimate will be estimated using a Relative Risk with 95% CI. ANOVA will be use for measures between the groups and along time, and correlation tests for anxiety and physical activity with gestational and perinatal variables.

DETAILED DESCRIPTION:
Participants, 192 nulliparous women that receive pre-natal care, allocated according to randomization into two groups: group one in which the women who participate in a program with physical and educational activities and the non-interventional group that will not receive the intervention and will follow a regular pre-natal care at routine of the service. The designation of participants will be performed, after informed consent will be sign, by opening sequentially envelopes previously sealed and numbered that will contain the information, previously generated by a computer system.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women aged between 16 and 40 years old
2. gestational age >20 weeks
3. nulliparous women
4. single fetus
5. Performing pre-natal care.

Exclusion Criteria:

1. Pathological heart condition
2. diabetes
3. hypertension
4. asthma bronchial
5. HIV+
6. gestational hypertension
7. gestational diabetes
8. pre-eclampsia
9. persistent bleeding
10. premature labor
11. cervical incompetence
12. acute infection with fever
13. restriction in fetal growth
14. indication of elective caesarian-section
15. in psychotherapy
16. performing other physical activity more than once a week.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 192 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-09 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
To assess the well being of the women trought the proportion of women with back pain and stress urinary incontinence | The outcome will be that the pregnant women will be interview at an average of up to 30 days after delivery
  To evaluate a well being in women who were receive intense care during prenatal care by the proportion of women with back pain and those with stress urinary incontinence

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Atençao Integral a Saude da Mulher CAISM, Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735
- [Derived] Miquelutti MA, Cecatti JG, Makuch MY. Developing strategies to be added to the protocol for antenatal care: an exercise and birth preparation program. Clinics (Sao Paulo). 2015 Apr;70(4):231-6. doi: 10.6061/clinics/2015(04)02. PMID 26017787
- [Derived] Miquelutti MA, Cecatti JG, Makuch MY. Antenatal education and the birthing experience of Brazilian women: a qualitative study. BMC Pregnancy Childbirth. 2013 Sep 5;13:171. doi: 10.1186/1471-2393-13-171. PMID 24007540
- [Derived] Miquelutti MA, Cecatti JG, Makuch MY. Evaluation of a birth preparation program on lumbopelvic pain, urinary incontinence, anxiety and exercise: a randomized controlled trial. BMC Pregnancy Childbirth. 2013 Jul 29;13:154. doi: 10.1186/1471-2393-13-154. PMID 23895188